CLINICAL TRIAL: NCT04564508
Title: Evaluation of Sodium Status in Septic and Septic Shock Patients and Its Relation to Prognosis and Hospital Stay
Brief Title: Sodium Status in Septic Patients and Its Relation to Prognosis an Hospital Stay
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kareem Sherif, Principal investigator, Assiut University
Other Study IDs: Sodium level in septic patient
Record Dates: First submitted 2020-09-21; First posted 2020-09-25 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Sodium Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The aim of the present study is to identify the prevalence and prognostic impact of sodium imbalance on sepsis and septic shock patients

DETAILED DESCRIPTION:
Sepsis and septic shock are among the most prevalent causes of intensive care unit (ICU) admissions. They account for around 10-50% of the mortality rate, which remains high despite extensive research of the Surviving Sepsis Campaign, and national core measures Sepsis is defined as "Organ dysfunction that threatens the patient's life caused by the impaired host response to infection" septic shock is defined as hypotension and serum lactate level greater than two mmol/L, as well as not responding to adequate fluid resuscitation requiring the use of vasopressors to maintain the mean blood pressure of 65 mm Hg or higher . Sepsis and septic shock are considered medical emergencies .

Acute hypernatremia is considered one of the features of homeostasis disturbances, which is common in septic patients with an incidence reaching up to 47% Finding biomarkers which predict the outcome of sepsis is challenging . Since electrolyte imbalance, specifically hypernatremia, is one of the commonest problems associated with sepsis and septic shock patients [20, 21]. It is, therefore, of current interest to study the evolution of sepsis in patients who have been shown to have hypernatremia.

Recent evidence shows that serum sodium levels may not be completely explained by fluid balance or sodium intake . Some studies suggest that sodium is intimately tied to the immune system, thus raising the question of whether inflammatory states such as sepsis can play a role in the development of hypernatremia

ELIGIBILITY:
Inclusion Criteria:

The diagnosis of sepsis and septic shock was made prior to the ICU admission. Sepsis and septic shock were defined according to the 3 definition using the Quick Sofa score of 2 or more

Sepsis : 2 or more of the SIRS criteria :

* Temperature >38 or <36 c
* Heart Rate >90 beats/minute
* Respiratory rate >20 cycle /minute
* wbc >20,000 or < 4,000 Plus the presumed existence of infection
* Blood pressure can be normal Septic shock : the same as sepsis plus refractory hypotension
* After bolus of 20- 40 ml/kg patient has one of the following :

  * SBP >90 mm Hg
  * MAP <65 mm Hg
  * Decrease of 40 mm Hg of base line hypernatremia [Na+]> 145 mmol/L eunatremia [135-145]mmol/l hyponatremia <135 mmol/L

Exclusion Criteria:

patients under the age of 18 years patients with a previous diagnosis of hyperaldosteronism patints diagnosed with Cushing syndrome, patients diagnosed with diabetes insipidus.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Septic and septic shock patients admitted to the ICU to evaluate their sodium status
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Sodium level disorders in Sepsis | Baseline
  Correlation between sodium level disorders in septic and septic shock patients and the outcome represented by ICU mortality and ICU length stay